CLINICAL TRIAL: NCT02068937
Title: Effectiveness of a Diuretic Algorithm in Clinical Stability and Readmissions in Heart Failure Patients
Brief Title: Effectiveness of a Diuretic Algorithm in Clinical Stability in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GPPG/HCPA 10-0376
Record Dates: First submitted 2014-02-17; First posted 2014-02-21 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Therapy; Diuretics; Algorithms
MeSH Terms: conditions — Heart Failure | interventions — Furosemide; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): In the control group, patients just diuretic adjusted (Furosemide 40 milligrams) by the doctor on the baseline. The patients do not receive phone calls neither advising on non-pharmacological treatment; The medication is adjusted by the doctor during the initial evaluation of study baseline.
  Interventions: Drug: Furosemide
- Furosemide and Phone contact (Experimental): The intervention group is conducted by a nurse in a systematic way during one time per week. If signs and symptoms of congestion, the dose of diuretic ( furosemide ) is revised , nonpharmacological guidelines are provided. According to the algorithm 1KG weight changes are indicative of modifying the diuretic dose , with the addition or reduction 1 tablet a day.
  Interventions: Drug: Furosemide and Phone contact

INTERVENTIONS:
Drug: Furosemide and Phone contact — The intervention group is conducted by a nurse in a systematic way during one time per week. If signs and symptoms of congestion, the dose of diuretic ( furosemide ) is revised , nonpharmacological guidelines are provided. According to the algorithm 1KG weight changes are indicative of modifying the diuretic dose , with the addition or reduction 1 tablet a day (1 tablet equivalent to 40 milligrams of furosemide)
  Other Names: phone calls
  Arms: Furosemide and Phone contact
Drug: Furosemide — This group received just diuretic adjusted (Furosemide 40 milligrams) by the doctor on the baseline.
  Other Names: Control Group
  Arms: Control Group

SUMMARY:
One of the challenges in treating patients with heart failure (HF) is achieving clinical stability and reducing the hospital readmission rate. A diuretic dose adjustment algorithm developed in the United States (Diuretic Treatment Algorithm, DTA) and later validated for use in Brazil (as the Algoritmo de Ajuste de Diurético, AAD) has proved feasible and readily applicable, but its effect on clinical outcomes has yet to be assessed. This report aims to describe a randomized clinical trial protocol designed to assess the effectiveness of the AAD and of nonpharmacologic management in improving clinical stability and reducing the readmission rate at 90 days in patients with HF.

DETAILED DESCRIPTION:
A PROBE (prospective randomized open blinded endpoint) parallel-group design will be used. Adult patients with a diagnosis of reduced ejection fraction HF, who are being treated at a specialized HF clinic are being recruited. Those with indications for loop diuretic dose adjustment during routine clinic visits will be randomized to take part in the trial. Participants in the intervention group (IG) shall have their diuretic doses adjusted in accordance with the AAD and receive four telephone calls (one per week) over 30 days to reinforce guidance on nonpharmacological management (fluid and sodium restriction). Participants in the control group (CG) shall have their diuretic doses adjusted by a physician during the first trial visit and shall not receive any telephone calls. Patients in both groups shall return at 1 month for face-to-face reassessment. The study endpoints shall comprise readmission and/or emergency department visits due to HF decompensation within 90 days and clinical instability. All participants shall be required to have a scale at home (or easy access to one), a telephone number, agree to telephone-based follow-up, and be available to return for a 1-month trial visit. Overall, 135 patients are expected to be enrolled in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* Age ≥ 18 years
* Diagnosed with systolic HF
* Able to monitor body weight at home
* Using furosemide

Exclusion Criteria:

* Those who are not able to make return visits or participate in telephone contact, and those on renal replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Compose outcome with readmission and/or emergency department visits due to HF decompensation within 90 days and clinical instability. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Eneida R Rabelo da Silva, ScD, Principal Investigator — HCPA and UFRGS
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Feijo MK, Ruschel KB, Bernardes D, Ferro EB, Rohde LE, Biolo A, Rabelo da Silva ER. Effects of a diuretic adjustment algorithm protocol on heart failure admissions: A randomized clinical trial. J Telemed Telecare. 2021 Jun;27(5):288-297. doi: 10.1177/1357633X211009640. Epub 2021 May 9. PMID 33966521
- [Derived] Feijo MK, Biolo A, Ruschel KB, Orlandin L, Aliti GB, Rabelo-Silva ER. Effect of a diuretic adjustment algorithm and nonpharmacologic management in patients with heart failure: study protocol for a randomized controlled trial. Trials. 2015 Feb 8;16:44. doi: 10.1186/s13063-015-0559-7. PMID 25885424